CLINICAL TRIAL: NCT01797328
Title: Study of the Effects of Temperature on Amount of Brown Adipose Tissue in Humans
Brief Title: Does Cold Provocation Increase Brown Adipose Tissue Volume?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Fredrik H Nystrom, Professor, MD, Head of internal medicine, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Nystrom_koldstudie; Dnr2013/41-32 (Other: Linkoping review board, Sweden)
Record Dates: First submitted 2013-02-18; First posted 2013-02-22 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Brown Adipose Tissue, Human
Keywords: brown adipose tissue, human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cold provocation (Active Comparator): cold arm
  Interventions: Procedure: cold arm
- to avoid feeling cold (Active Comparator): warm arm
  Interventions: Procedure: warm arm

INTERVENTIONS:
Procedure: cold arm — 1 hour/day of cold provocation of such an extent that it is unpleasant but does not cause shivering
  Arms: cold provocation
Procedure: warm arm — To the best of ability avoid feeling cold during 6 weeks
  Arms: to avoid feeling cold

SUMMARY:
About 28 healthy subjects are randomized to 1 hour/day of coldprovocation or to the best of ability to avoid feeling cold, for 6 weeks. Basal metabolic rate and magnetic resonance (for determination of brown adipose tissue volume) imaging are performed before and after the study.

ELIGIBILITY:
Inclusion Criteria: healthy subjects -

Exclusion Criteria: any significant disease, ot other conditions that interferes with magnetic resonance imaging

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-02; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Science, Linköping, Linköping, Sweden

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cold Provocation | to Avoid Feeling Cold
Started | 16 | 12
Completed | 14 | 12
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: Healthy non-obese subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Cold Provocation | to Avoid Feeling Cold | Total
Number analyzed (Participants) | 16 | 12 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 12 | 28
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Continuous data was only available for those 14 participants who completed the study Population: because there were 14 who did the study
  years
    number analyzed (Participants) | 14 | 12 | 26
    (all) | 26.1 (3.9) | 24.3 (2.9) | 25.3 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: because 2 did not do the study at all
  Participants
    number analyzed (Participants) | 14 | 12 | 26
    Female | 9 | 7 | 16
    Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  Sweden | 16 | 12 | 28

OUTCOME MEASURES:

1. Primary Outcome: Brown Adipose Tissue, Absolute Volume
Description: Sub-clavicular brown adipose tissue volume by magnetic resonance imaging (liters)
Time Frame: Baseline and 6 week
Population: Brown adipose tissue volume (liters)
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Cold Provocation | to Avoid Feeling Cold
Number analyzed (Participants) | 13 | 12
liters | 0.0066 (0.012) | 0.0021 (0.0086)

ADVERSE EVENTS:
Groups:
- Cold Provocation: cold arm
  cold arm: 1 hour/day of cold provocation of such an extent that it is unpleasant but does not cause shivering
  no reported adverse events
Arm/Group | Cold Provocation | to Avoid Feeling Cold
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/12
Other Adverse Events (participants affected / at risk) | 0/16 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No